CLINICAL TRIAL: NCT05884125
Title: Promoting Healing of Injured Nerves With Electrical Stimulation Therapy
Acronym: PHINEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Checkpoint Surgical Inc. (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0153-CSP-002; W81XWH1920065 (Other Grant/Funding Number: Department of Defense USAMRAA)
Record Dates: First submitted 2023-05-19; First posted 2023-06-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Nerve Injury; Peripheral Nerve Injuries; Peripheral Nerve Injury Upper Limb; Nerve Palsy
Keywords: Therapeutic Electrical Stimulation; Brief Electrical Stimulation; Nerve Regeneration; Nerve Injury; Nerve Healing; Nerve Repair
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Brief Electrical Stimulation Therapy (Experimental): Single, 10 minute dose of electrical stimulation delivered to the injured nerve during surgical intervention.
  Interventions: Device: Checkpoint BEST System
- Standard of Care (No Intervention): Surgical intervention for repair of peripheral nerve injury.

INTERVENTIONS:
Device: Checkpoint BEST System — Single use medical device, consisting of electric stimulator and intraoperative lead. Therapy consists of single, 10 minute dose delivered proximal to site of decompression/repair
  Other Names: Brief Electrical Stimulation (BES) Therapy
  Arms: Brief Electrical Stimulation Therapy

SUMMARY:
This study is evaluating a new therapeutic use of electrical stimulation to promote nerve healing and improve functional recovery following surgical intervention for peripheral nerve injury in arm. Participants will be randomized into one of two groups, treatment or control, with all participants receiving standard of care treatment for the nerve injury. The treatment group will also receive a single dose of the therapeutic stimulation during the surgical intervention for their nerve injury.

DETAILED DESCRIPTION:
Preliminary research has shown that delivering a brief period of electrical stimulation following nerve repair promotes nerve healing and functional recovery. This pilot study is investigating the use of a single dose of therapeutic electrical stimulation to promote nerve healing. The therapy is delivered as part of the surgical intervention to address peripheral nerve injury in the arm.

ELIGIBILITY:
Inclusion Criteria:

* Upper extremity mixed or motor nerve injury from the brachial plexus to the wrist crease.
* Candidate for surgical intervention.
* Indicated for surgical repair by nerve transfer, primary repair, or nerve grafting.
* Are age 18-80 years.
* Signed and dated informed consent form.

Exclusion Criteria:

* Severe comorbid condition, such as arrhythmia or congestive heart failure, preventing surgery.
* Primary repair requiring graft >6cm.
* Nerve reconstruction occurring >12 months post injury.
* Age less than 18 or greater than 80 years.
* All contraindications to included/required surgical procedure, including but not limited to language barriers, mental status barriers, inability to consent, and pregnancy/lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Motor Recovery assessed using the Medical Research Council (MRC) motor grading | Pre-surgery, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Grading of muscle strength on 0 to 5 scale, with higher score representing greater function.

SECONDARY OUTCOMES:
Grip Strength | Pre-surgery, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Maximum grip strength.
Lateral Pinch Strength | Pre-surgery, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Maximum lateral pinch.
2-point discrimination | Pre-surgery, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Evaluation of sensory function, measuring tactile discrimination.
Semmes-Weinstein Monofilament Testing | Pre-surgery, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Evaluation of sensory function, measuring pressure detection threshold.
Patient Reported Outcome Measurement System (PROMIS) Upper Extremity Function | Pre-surgery, 10 days, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Questionnaire providing patient reported estimate of upper extremity function on a 0-100 scale with >50 representing greater normal function.
Patient Reported Outcome Measurement System (PROMIS) Pain Interference | Pre-surgery, 10 days, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Questionnaire providing patient reported estimate of interference of pain on daily activities on a 0-100 scale with >50 representing greater than normal pain interference on daily activities.
quick Disabilities of thee Arm, Shoulder, and Hand (DASH) questionnaire | Pre-surgery, 10 days, 2 months, 4 months, 6 months, 8 months, 10 months, 12 months, 15 months, and 18 months
  Questionnaire providing patient reported estimate upper extremity function. The score ranges from 0 (no disability) to 100 (most severe disability).
Electromyography (EMG) | 4 months, 6 months, and 8 months
  Measurement of the electrical activity in a muscle.
Motor Unit Number Estimation (MUNE) | 4 months, 6 months, and 8 months
  Estimate of the number of motor units within the muscle based on recorded electrical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Moore, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Univeristy - Department of Plastic and Reconstructive Surgery, Columbus, Ohio, United States

REFERENCES:
- [Background] Jo S, Pan D, Halevi AE, Roh J, Schellhardt L, Hunter Ra DA, Snyder-Warwick AK, Moore AM, Mackinnon SE, Wood MD. Comparing electrical stimulation and tacrolimus (FK506) to enhance treating nerve injuries. Muscle Nerve. 2019 Nov;60(5):629-636. doi: 10.1002/mus.26659. Epub 2019 Aug 21. PMID 31397919
- [Background] Sayanagi J, Acevedo-Cintron JA, Pan D, Schellhardt L, Hunter DA, Snyder-Warwick AK, Mackinnon SE, Wood MD. Brief Electrical Stimulation Accelerates Axon Regeneration and Promotes Recovery Following Nerve Transection and Repair in Mice. J Bone Joint Surg Am. 2021 Oct 20;103(20):e80. doi: 10.2106/JBJS.20.01965. PMID 34668879
- [Background] Roh J, Schellhardt L, Keane GC, Hunter DA, Moore AM, Snyder-Warwick AK, Mackinnon SE, Wood MD. Short-Duration, Pulsatile, Electrical Stimulation Therapy Accelerates Axon Regeneration and Recovery following Tibial Nerve Injury and Repair in Rats. Plast Reconstr Surg. 2022 Apr 1;149(4):681e-690e. doi: 10.1097/PRS.0000000000008924. PMID 35139047
- [Background] Wong JN, Olson JL, Morhart MJ, Chan KM. Electrical stimulation enhances sensory recovery: a randomized controlled trial. Ann Neurol. 2015 Jun;77(6):996-1006. doi: 10.1002/ana.24397. Epub 2015 May 4. PMID 25727139
- [Background] Juckett L, Saffari TM, Ormseth B, Senger JL, Moore AM. The Effect of Electrical Stimulation on Nerve Regeneration Following Peripheral Nerve Injury. Biomolecules. 2022 Dec 12;12(12):1856. doi: 10.3390/biom12121856. PMID 36551285
- [Background] Keane GC, Pan D, Roh J, Larson EL, Schellhardt L, Hunter DA, Snyder-Warwick AK, Moore AM, Mackinnon SE, Wood MD. The Effects of Intraoperative Electrical Stimulation on Regeneration and Recovery After Nerve Isograft Repair in a Rat Model. Hand (N Y). 2022 May;17(3):540-548. doi: 10.1177/1558944720939200. Epub 2020 Jul 15. PMID 32666827